CLINICAL TRIAL: NCT07212465
Title: Feasibility, Tolerability, and Preliminary Efficacy for Non-Invasive Neuromodulation of the Anterior Cingulate Cortex for Depression (NACC-D) in Older Adults Using Deep Transcranial Magnetic Stimulation With an Accelerated Intermittent Theta Burst Protocol
Brief Title: Accelerated Neuromodulation of Anterior Cingulate Cortex for Depression
Acronym: NACC-D
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rotman Research Institute at Baycrest (Other)
Responsible Party: Principal Investigator, Linda Mah, MD, Clinician Scientist, Rotman Research Institute at Baycrest
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 25-03
Record Dates: First submitted 2025-09-11; First posted 2025-10-08 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-09

CONDITIONS: Major Depressive Disorder (MDD)
Keywords: Transcranial Magnetic Stimulation (TMS); Treatment Resistant Depression; Intermittent Theta Burst Stimulation
MeSH Terms: conditions — Depressive Disorder, Major; Depressive Disorder, Treatment-Resistant

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- 20-40 sessions of sham stimulation (Sham Comparator): Participants will receive sham intervention if randomized into sham condition. The sham intervention consists of treatment with similar technical parameters which induce scalp sensations but do not penetrate into the brain.
  Interventions: Device: Sham Brainsway H1-Coil Deep TMS System
- 20-40 sessions of iTBS dTMS (Experimental): Participants will receive dTMS if randomized into the active condition. The motor threshold (MT) will be measured by delivering single stimulations to the motor cortex with gradually increased intensity. The stimulation protocol consists of 6-8 dTMS sessions of intermittent theta burst stimulation delivered at an intensity of 80-90% of resting MT each day for five consecutive days
  Interventions: Device: Active Brainsway H7-Coil Deep TMS System

INTERVENTIONS:
Device: Active Brainsway H7-Coil Deep TMS System — Deep Transcranial Magnetic Stimulation (dTMS) is a new form of TMS which allows direct stimulation of deeper neuronal pathways than the standard TMS. The H-coil is a novel dTMS coil designed to allow deeper brain stimulation without a significant increase of electric fields induced in superficial cortical regions. dTMS will be administered 6-8 times a day for 5 consecutive days.
  Arms: 20-40 sessions of iTBS dTMS
Device: Sham Brainsway H1-Coil Deep TMS System — In addition to the active H7-coil, a sham coil is included in the H1-coil helmet. The sham treatment will be administered 6-8 times a day for 5 consecutive days.
  Arms: 20-40 sessions of sham stimulation

SUMMARY:
The goal of this clinical trial is to test whether an accelerated deep Transcranial Magnetic Stimulation (dTMS) protocol can reduce depressive symptoms in older adults (ages 60-85) with Major Depressive Disorder (MDD) who have not tolerated or responded to antidepressant medications. The study will evaluate whether accelerated dTMS administered over 5 consecutive days is safe and well-tolerated in this population, and whether it produces greater reductions in depressive symptoms compared to placebo stimulation.

DETAILED DESCRIPTION:
This study will investigate the effects of an accelerated intermittent theta burst protocol (a-iTBS) using the H7 deep Transcranial Magnetic Stimulation (dTMS) coil to target the anterior cingulate cortex (ACC) in older adults (aged 60-85) with Major Depressive Disorder (MDD). Twenty-four older adults with treatment-resistant MDD will participate in a single site, double-blind, randomized sham-controlled trial using an accelerated schedule of multiple dTMS sessions per day for 5 consecutive days. The primary goal of the study is to establish the feasibility of an accelerated aiTBS protocol of the ACC in older adults with treatment resistant depression, and to obtain preliminary evidence of treatment efficacy.

ELIGIBILITY:
Inclusion Criteria:

* are between 60- 85 years old (on the day of randomization)
* have been diagnosed with DSM5 Major Depressive Disorder, with the current episode longer than 4 weeks but less than 5 years
* did not respond to/did not tolerate, or failed to achieve remission with at least one antidepressant trial of 8 week minimum duration
* are willing to provide informed consent
* are able to follow the treatment schedule
* are stable on medications for 2 months and are not expected to change medication during the entire study period (if they are taking medications)
* have a satisfactory safety screening questionnaire for TMS

Exclusion Criteria:

* have a metal plate in your head (such as an ear implant, implanted brain stimulators, aneurysm clips). Dental devices and implants that are non-magnetic are safe
* have known increased pressure or a history of increased pressure in their brain, which may increase their risk for having seizures
* have a cardiac pacemaker
* have an implanted medication pump
* have a central venous line
* have a history of any psychotic disorder, bipolar disorder, eating disorder, obsessive compulsive disorder, post-traumatic stress disorder, or dementia
* have a history of substance abuse in the last 6 months
* have a history of stroke or other brain lesions
* have a personal history of epilepsy
* have a family history of epilepsy
* are a pregnant or breast-feeding woman
* have a history of abnormal MRI of the brain
* have untreated hypo- or hyper-thyroidism
* have unstable medical condition(s)
* have any other known contraindications to TMS
* are on unstable doses of any psychotropic medication such as - antidepressants, antipsychotic, mood stabilizers or memory enhancing medications
* require daily doses of benzodiazepines or hypnotics within two weeks of randomization

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-07-21 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-02-15 (Estimated)

PRIMARY OUTCOMES:
Percentage of scheduled treatment sessions that are attended by study participants | 6 weeks
Participant-reported comfort and feasibility based on the frequency and type of adverse events as measured using the Adverse Events Questionnaire (AEQ) | 6 weeks
  Severity of symptoms is rated from 1 to 4, with 1 being absent and 4 being severe. Whether symptoms are perceived to be relatedTMS treatment are rated from 1 to 5, with 1 being no and 5 being definitely.
The number of participants who have prematurely withdraw and reasons for withdrawal | 6 weeks
The change from baseline in Montgomery-Asberg Depression Rating Scale (MADRS) scores following the final treatment on day 5 (i.e., after 5 days of H7-coil a-iTBS) in the treatment group compared to the sham group. | 1 week
  An effect size (Cohen's d) of 0.5 will be considered a minimally important effective size. The MADRS ranges from 0-60, with a greater score indicating greater depressive symptoms.

SECONDARY OUTCOMES:
Response rates compared between treatment groups following 5 days of treatment, where the response rate refers to the percentage of patients who responded to a-ITBS treatment and response is defined as a ≥50% reduction in MADRS score from baseline | 6 weeks
  Response rates will be compared from baseline to after 5 day treatment and at 1 month follow-up. MADRS scores range from 0-60, with a greater score indicating greater severity of depressive symptoms.
Remission rates compared between treatment groups following 5 days of treatment, where the remission rate is defined as MADRS score <10 | 6 weeks
  MADRS scores will be compared between baseline, after 5 days of treatment and at 1-month follow-up. The MADRS ranges from 0-60, with a greater score indicating greater depressive symptoms
The change in baseline slow wave and resting state activity as measured with electroencephalography (EEG) following 5 days of treatment and at 1-month follow-up | 6 weeks
The change in functional connectivity within the default mode and central autonomic networks on Magnetic Resonance Imaging (MRI) | 1 week
The change in slow wave activity in the posterior default mode network (posterior cingulate cortex) as measured with MEG | 1 week
The change in baseline cognitive tests following 5 days of treatment and at 1-month follow-up (cognitive domains tested include executive function and memory), | 6 weeks
  Baseline cognitive tests will be measured using a neuropsychological test battery.
The change in baseline resting state heart rate variability (HRV) following a single TMS session and after 5 days of treatment | 1 week
The change in baseline emotional processing as measured with an Affective Simon task following a single TMS session, after 5 days of treatment and at 1-month follow-up | 6 weeks
  The Affective Simon task will measure the number of correct responses to stimuli in the task.

CONTACTS AND LOCATIONS:
Overall Officials: Linda Mah, MD, Principal Investigator — Baycrest Rotman Research Institute
Locations (1):
- Rotman Research Institute at Baycrest, Toronto, Ontario, Canada